CLINICAL TRIAL: NCT06575010
Title: Single-Shot Liposomal Bupivacaine vs. Liposomal Bupivacaine Combined With Dexamethasone Following Arthroscopic Rotator Cuff Repair: A Prospective Randomized Controlled Trial
Brief Title: Exparel v Dexamethasone in RCR
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0726SNAM
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Rotator Cuff Tears; Postoperative Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Shoulder Block using Exparel (Active Comparator): Participants having rotator cuff repair surgery will receive Liposomal bupivacaine (Exparel) + bupivacaine given in their shoulder block before surgery.
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine Hcl 0.5% Inj
- Group 2: Shoulder Block using Exparel + Dexamethasone (Active Comparator): Participants having rotator cuff repair surgery will receive Liposomal bupivacaine (Exparel) + Dexamethasone + bupivacaine given in their shoulder block before surgery.
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine Hcl 0.5% Inj; Drug: Dexamethasone

INTERVENTIONS:
Drug: Liposomal bupivacaine — 20 mL Liposomal bupivacaine (Exparel) will be given in the shoulder block prior to surgery
Drug: Bupivacaine Hcl 0.5% Inj — 0.75% bupivacaine will be given in the shoulder block prior to surgery
Drug: Dexamethasone — 10 mg Dexamethasone will be given in the shoulder block prior to surgery
  Arms: Group 2: Shoulder Block using Exparel + Dexamethasone

SUMMARY:
Effective and safe control of pain after shoulder surgery is an important component of the post-surgical process. Patients who are comfortable in the early period after surgery are more satisfied with their experience and are better able to participate in rehabilitation exercises during their stay in the hospital. As surgeons and health care systems in the United States find themselves in the middle of an opioid epidemic, it is necessary to discover different options to provide patients pain relief that are both effective and safe in an effort to decrease the amount of pain medication used.

ELIGIBILITY:
Inclusion Criteria:

* Participants having a primary rotator cuff repair
* Age 18 and older
* English speaking
* Ability to complete surveys by phone or in person
* Ability to provide informed consent

Exclusion Criteria:

* Revision rotator cuff repair (RCR) cases
* Participants having an open RCR
* Allergies and/or medical contra-indications to study medications
* Non-English speakers
* Participants who are pregnant, plan to become pregnant and do not utilize adequate contraceptive means, or are currently breastfeeding (all patients who have the potential to be pregnant are administered a urine beta-HCG pregnancy test, with suspected false-positive or equivocal urine pregnancy tests followed by a more specific serum pregnancy test)
* Rotator cuff repair needing Graft Augmentation
* Known alcohol or narcotic abuse history
* Existing contract with a pain specialist due to underlying preoperative pain syndrome
* Preoperative opioid use within the 3 months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-08-26 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative narcotic medication use | 14 days
  Participants will be asked to record the amount of medication they take to control pain after surgery
Postoperative pain levels | 14 days
  This will be measured by providing participants the visual analog scale (VAS) questionnaire as well as a postoperative pain recording diary to complete after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States